CLINICAL TRIAL: NCT01910974
Title: TRESTIS: Multicentric Study With a Curative Endoscopic Treatment of Superficial Neoplasia of a Digestive Tract by Endoscopic Submucosal Dissection: Evaluation of a New Water Jet System Injecting Glycerol Mix
Brief Title: Multicentric Study an Endoscopic Treatment of Digestive Neoplasia by Submucosal Dissection Evaluation of a New Water Jet System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Edouard Herriot (Other)
Responsible Party: Principal Investigator, Jean Christophe Saurin, Thieery Ponchon, Hôpital Edouard Herriot
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRESTIS 2013-A00133-42; TRESTIS (Other: RCB 2013-A00133-42)
Record Dates: First submitted 2013-07-15; First posted 2013-07-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2012-07

CONDITIONS: Stomach Neoplasm; Intestinal Neoplasm; Rectal Neoplasm
Keywords: oesophagus; stomach; intestine; rectum
MeSH Terms: conditions — Stomach Neoplasms; Intestinal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- endoscopic sub-mucosal dissection (Experimental)
  Interventions: Procedure: endoscopic sub-mucosal dissection

INTERVENTIONS:
Procedure: endoscopic sub-mucosal dissection — endoscopic sub mucosal dissection of oesophagus stomach intestine or rectum lesions

SUMMARY:
safety evaluation of endoscopic sub-mucosal dissection with nestis enki2 system. This system is a new water jet system which allows to perform Endoscopic submucosal dissection with a bifunctional catheter (injection and cutting).

DETAILED DESCRIPTION:
Evaluation of the ability of this system to have a complete resection of superficial tumors of the digestive tract (that is to say a resection with free lateral and deep margins without residual tumor tissue)

Evaluation of the ability of such system to inject a viscous macromolecular solution of glycerol (glycerol mix: Glycerol 10 %, Fructose 5 %, saline solution 0.9%)(27. Fujishiro M, Yahagi N, Kashimura K, et al. Comparison of various submucosal injection solutions for maintaining mucosal elevation during endoscopic mucosal resection. Endoscopy. 2004;36:579-583.)

ELIGIBILITY:
Inclusion Criteria:

* OVER 18 YEARS OLD
* PATIENTS AGREED WITH THE STUDY
* SCORE ASA 1 OR 2
* Patient recorded in a social safety organism
* patients presenting with superficial lesions with an endoscopic indication of resection

Exclusion Criteria:

* under 18 years old
* Patients not agreed with the study
* pregnant women
* patient included in an another study
* medical treatments (radiotherapy, surgery endoscopis treatements) before the intervention
* coagulation disorders
* score asa over 3
* patients with another neoplasic lesion

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
SAFETY THAT IS TO SAY PERFORATION RATE AND delayed BLEEDING ONE | 18 months
  inclusion duration is about 6 months the following period will be about 12 months so a total duration of 18 months

CONTACTS AND LOCATIONS:
Overall Officials: PINSET CHRISTIAN, CEO, Study Director — SPONSOR DIRECTOR
Locations (1):
- NESTIS, Lyon, Auvergne-Rhône-Alpes, France